CLINICAL TRIAL: NCT07279623
Title: Intra-Nasal Mechanical Stimulation (INMEST) as a Potential Preventative Treatment for Migraine - A Prospective, Randomized, Open Label, Delayed-Start Study to Evaluate the Safety and Performance of the Walther System
Brief Title: Intra-Nasal Mechanical Stimulation (INMEST) as a Potential Preventative Treatment for Migraine
Acronym: A-MI-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abilion Medical Systems AB (Industry)
Collaborators: Aurevia (Industry); Insamlingsstiftelsen för främjande av forskning avseende INMEST (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-MI-01; CIV-25-05-052936 (Registry Identifier: Swedish Clinical Trials Registry)
Record Dates: First submitted 2025-11-18; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: Migraine
Keywords: Migraine; Migraine prophylaxis / Preventive treatment; Neuromodulation; Intra-nasal mechanical stimulation; INMEST; Medical device; Chronic migraine; Episodic migraine; Headache disorders
MeSH Terms: conditions — Migraine Disorders; Headache Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Early Start (Active Comparator): Subjects undergo a 4-week baseline assessment (weeks 1-4), then receive active treatment with the Walther System every second day for 6 weeks (weeks 5-10). The first treatment is performed under supervision at the clinic, and subsequent treatments are self-administered at home. Post-treatment assessments occur during weeks 11-14.
  Interventions: Device: INMEST-treatment
- Group B - Delayed Start (Active Comparator): Subjects undergo a 4-week baseline assessment (weeks 1-4), followed by a 6-week no-treatment reference period (weeks 5-10). Active treatment with the Walther System is then administered every second day for 6 weeks (weeks 11-16), starting with an initial supervised treatment at the clinic. Post-treatment assessments occur during weeks 17-20.
  Interventions: Device: INMEST-treatment

INTERVENTIONS:
Device: INMEST-treatment — Hand-held controller and catheter assembly for intra-nasal mechanical stimulation (INMEST), self-administered at home every second day for 6 weeks, first treatment under supervision.
  Other Names: Walther System

SUMMARY:
This is a prospective, randomized, open-label, delayed-start clinical investigation evaluating the safety and efficacy of the Walther System, a Class IIa investigational medical device delivering intra-nasal mechanical stimulation (INMEST), as a preventative treatment for migraine. A total of 110 adults (18-65 years) with a history of migraine will be randomized 1:1 into two groups: Group A (early treatment) and Group B (delayed treatment). The study includes baseline assessments, in-clinic device training, and home-based self-administered treatments every second day for six weeks. The primary outcome is the change in monthly migraine days during the primary treatment comparison period. Secondary outcomes include headache days, migraine intensity, duration, rescue medication use, patient-reported outcomes, device compliance, and safety. The study will be conducted at one site in Sweden.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years at the time of screening.
2. The study subject must have a clinical diagnosis of migraine without aura, migraine with aura, or chronic migraine according to the 3rd edition of the International Classification of Headache Disorder (ICHD-3), indicated by medical record shown by the subject.
3. Onset of migraine headache occurred before age 50.
4. History of migraines for at least 1 year before screening.
5. The study subject reports at least 8 monthly migraine days during the screening period.
6. If subject is on a prophylactic migraine medication regimen:

   1. Reports stable medication regimen during the three months prior to screening.
   2. Able and willing to maintain medication regimen (no change in type, frequency or dose) from screening to end of follow-up.
7. The study subject reports having understood and have signed the Informed Consent Form (ICF) and is willing to comply with all investigation visits and assessments.
8. Women of childbearing potential must agree to use a reliable, medically approved form of contraception during the study participation until end of study.
9. Anticipated compliance with prescribed treatment and follow-up.

Exclusion Criteria:

1. Subject unable to distinguish between migraine headaches and other headache types.
2. Recently (12 months prior screening) undergone nasal or sinus surgery.
3. Any severe diseases for which, in the opinion of the Investigator, participation would not be in the best interest of the subject or that can interfere with the performance, evaluation, and outcome of the clinical evaluation.
4. Previous (within 30 days prior to screening) and concurrent treatment with another investigational drug/s or device/s.
5. Subject is pregnant or lactating or planning to get pregnant during the duration of the study.
6. The study subject has a cognitive incapacity or language barrier precluding adequate understanding or cooperation.
7. The study subject is considered by the Investigator to be unsuitable to participate in the investigation for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Monthly Migraine Days | Weeks 7-10 (Group A: Treatment performance period; Group B: No treatment reference period)
  Between-group comparison of the difference in mean change in monthly migraine days from the baseline assessment period (weeks 1-4) to Group A) Treatment performance period (weeks 7-10) and Group B) No treatment reference period (weeks 7-10).

SECONDARY OUTCOMES:
Mean change in monthly headache days | Weeks 7-10
  Between-group comparison of the difference in mean change in monthly headache days from baseline.
Mean change in migraine intensity | Weeks 7-10
  Between-group comparison of the difference in mean change in migraine intensity from baseline.
Mean change in duration of migraine attacks | Weeks 7-10
  Between-group comparison of the difference in mean change in migraine attack duration (hours) from baseline.
Proportion of attacks requiring rescue medication | Weeks 7-10
  Between-group comparison of the proportion of migraine attacks requiring rescue medication.
Number of participants with ≥30% and ≥50% reduction in monthly migraine days | Weeks 7-10
  Between-group comparison of the proportion of subjects achieving ≥30% and ≥50% reduction in monthly migraine days.
Mean change in PROMIS-PI SF-6b | Weeks 7-10
  Between-group comparison of the difference in mean change from baseline in PROMIS-PI SF-6b scores. The raw scores are converted to standardized T-scores (range 0-100; mean = 50, SD = 10) based on the PROMIS calibration sample. Higher scores indicate greater pain-related interference.
Mean change in Migraine-Specific Quality of Life Questionnaire (MSQ) | Weeks 7-10
  Between-group comparison of the difference in mean change from baseline in MSQ scores. Scores are transformed to a 0-100 scale, with higher scores indicating better quality of life.
Mean change in Patient Global Impression of Severity (PGI-S) | Weeks 7-10
  Between-group comparison of the difference in mean change from baseline in PGI-S scores. Measured on a 7-point scale (1 = least severe, 7 = most severe), where higher values indicate greater severity.
Mean change in monthly migraine days | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in monthly migraine days within each group.
Mean change in monthly headache days | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in monthly headache days within each group.
Mean change in migraine intensity (6-point severity scale) | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in migraine intensity within each group. Migraine intensity is assessed using a 6-point severity scale (1 = Very mild, 6 = Very severe), where higher scores indicate greater pain severity.
Mean change in duration of migraine attacks | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in duration of migraine attacks (hours) within each group.
Proportion of migraine attacks requiring rescue medication | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Proportion of migraine attacks requiring rescue medication within each group.
Number of participants with ≥30% and ≥50% reduction in monthly migraine days | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Proportion of subjects achieving ≥30% and ≥50% reduction in monthly migraine days within each group.
Mean change in PROMIS-PI SF-6b | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in PROMIS-PI SF-6b scores within each group. The raw scores are converted to standardized T-scores (mean = 50, SD = 10) based on the PROMIS calibration sample. Higher scores indicate greater pain-related interference.
Mean change in Migraine-Specific Quality of Life Questionnaire (MSQ) | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in PROMIS-PI SF-6b, MSQ, and PGI-S scores within each group. Scores are transformed to a 0-100 scale, with higher scores indicating better quality of life.
Mean change in Patient Global Impression of Severity (PGI-S) | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in PGI-S scores within each group. Measured on a 7-point scale (1 = least severe, 7 = most severe), where higher values indicate greater severity.
Mean change in monthly migraine days | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in monthly migraine days, pooled across both groups.
Mean change in monthly headache days | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in monthly headache days, pooled across both groups.
Mean change in migraine intensity (6-point severity scale) | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in migraine intensity, pooled across both groups. Migraine intensity is assessed using a 6-point severity scale (1 = Very mild, 6 = Very severe), where higher scores indicate greater pain severity."
Mean change in duration of migraine attacks | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in duration of migraine attacks (hours), pooled across both groups.
Proportion of migraine attacks requiring rescue medication | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Proportion of migraine attacks requiring rescue medication, pooled across both groups.
Number of participants with ≥30% and ≥50% reduction in monthly migraine days | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Proportion of subjects achieving ≥30% and ≥50% reduction in monthly migraine days, pooled across both groups.
Mean change in PROMIS-PI SF-6b | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in PROMIS-PI SF-6b scores, pooled across both groups. The raw scores are converted to standardized T-scores (mean = 50, SD = 10) based on the PROMIS calibration sample. Higher scores indicate greater pain-related interference.
Mean change in Migraine-Specific Quality of Life Questionnaire (MSQ) | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in PROMIS-PI SF-6b, MSQ, and PGI-S scores, pooled across both groups. Scores are transformed to a 0-100 scale, with higher scores indicating better quality of life.
Mean change in Patient Global Impression of Severity (PGI-S) | Group A: Weeks 1-4 → 11-14; Group B: Weeks 7-10 → 17-20
  Change from baseline in PGI-S scores, pooled across both groups. Measured on a 7-point scale (1 = least severe, 7 = most severe), where higher values indicate greater severity.
Proportion of prescribed treatments completed | Throughout the 6-week treatment period
  Compliance based on device usage logs or participant-reported treatment diaries.
Adverse Events / Serious Adverse Events / Device Effects | Through study completion (14 or 20 weeks, depending on treatment group)
  Number of treatment-related AEs, SAEs, ADEs, SADEs, and Unanticipated SADEs for the Walther System.
Device Deficiencies | Throughout the 6-week treatment period
  Number of device deficiencies for the Walther System.

OTHER OUTCOMES:
Device usability and user experience (combined questionnaires) | Throughout the 6-week treatment period
  User-reported usability, ease of use, handling, and overall experience of the device during home use, assessed using two Device Usability Questionnaires. Questions include multiple 3- or 5-point scales, 0-10 scales, and yes/no responses. Higher scores indicate better usability or greater interest where applicable.
Symptom trends (Symptom Questionnaire) | Throughout the 6-week treatment period
  Changes in symptoms potentially related to autonomic nervous system function, assessed using the Symptom Questionnaire at Visits 1-5. The questionnaire includes multiple items with 0-6 and 0-3 ordinal scales, yes/no responses, and other response formats. Higher scores indicate more severe symptoms."

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Erik Juto, PhD, MD, Principal Investigator
Locations (1):
- INMEST-mottagningen Odenplan, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No